CLINICAL TRIAL: NCT02206841
Title: Establishment of Non-alcoholic Fatty Liver Disease Cohort and Development of Markers to Predict Histologic Progression of Liver Fibrosis
Brief Title: Establishment of NAFLD Cohort and Development of Fibrosis Markers
Acronym: NAFLD
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Boramae Hospital (Other)
Responsible Party: Principal Investigator, Won Kim, M.D, PhD, Seoul National University Boramae Hospital
Other Study IDs: NAFLD_cohort
Record Dates: First submitted 2014-07-28; First posted 2014-08-01 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Fibrosis of Liver
Keywords: fibrosis; markers
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Obtained blood samples will be stored by serum and plasma for future analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NAFLD: Patients with suspected nonalcoholic fatty liver disease will be screened. Of all patients fulfilling inclusion criteria, baseline characteristics will be obtained. In addition, laboratory, radiologic evaluations such as ARFI, SWE, and transient elastography will be performed. A diagnostic liver biopsy will be performed for analysis of steatosis and fibrosis. Parts of the remaining liver tissue will be stored by frozen tissue and paraffin block for future study. Several serum and plasma samples are collected of patients and stored for future analysis such as targeted SNP arrays, super-enhancer RNA (eRNA) expression, whole exome sequencing, RNA chip sequencing, RNA microarray, genomic DNA, metabolomics, fecal microbiome, metabolite, metagenome/metatranscriptome analyses.
  Interventions: Procedure: Liver biopsy; Device: ARFI; Device: SWE; Device: Transient elastography

INTERVENTIONS:
Procedure: Liver biopsy — Percutaneously liver biopsy will be performed for evaluate steatosis and fibrosis.
Device: ARFI — Acoustic radiation force impulse (ARFI) imaging will be performed for evaluate fibrosis of liver.
Device: SWE — Supersonic shear wave elastography (SWE) will be performed for evaluate fibrosis of liver.
Device: Transient elastography — Transient elastography will be performed for evaluate fibrosis of liver.

SUMMARY:
This study is designed for establishment of non-alcoholic fatty liver disease patients cohort to development of markers to predict histologic progression of liver fibrosis.

DETAILED DESCRIPTION:
* Acoustic radiation force impulse elastography and transient elastography
* Liver tissue (frozen tissue, paraffin block)
* Whole blood, Serum
* Fat amount ratio CT (Visceral adipose tissue, Subcutaneous adipose tissue amount)
* Body composition analyzer (InBody scale):Total fat/muscle mass and appendicular skeletal muscle mass
* Pulmonary function test with post-bronchodilator response and DLCo
* EKG, EchoCG, Heart CT (Coronary calcium score), and Pusle wave velocity (AI index, arterial stiffness)
* Brain MRI or CT
* Upper esophagogastroscopy and colonoscopy
* Berlin score questionnaire and Polysomnography

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed fatty liver disease
* Patients with radiologically confirmed fatty liver disease

Exclusion Criteria:

* History of significant alcohol consumption
* Viral hepatitis
* Autoimmune hepatitis
* Metabolic diseases (e.g. hemochromatosis, M. Wilson, alpha 1-antitrypsin deficiency)
* Hepatotoxic medication (e.g. amiodarone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-alcoholic fatty liver disease
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-01-01; Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
histologic steatosis and fibrosis grade | baseline
  We will evaluate fibrosis using laboratory examination, radiologic evaluation and liver tissue pathology.

SECONDARY OUTCOMES:
Development of markers for hepatic fibrosis progression | baseline and every 6 months (up to 1year)
  We will analysis and development fibrosis markers by obtained blood sample and liver tissue,

CONTACTS AND LOCATIONS:
Overall Officials: Won Kim, Professor, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koo BK, Joo SK, Kim D, Bae JM, Park JH, Kim JH, Kim W. Additive effects of PNPLA3 and TM6SF2 on the histological severity of non-alcoholic fatty liver disease. J Gastroenterol Hepatol. 2018 Jun;33(6):1277-1285. doi: 10.1111/jgh.14056. Epub 2018 Feb 26. PMID 29193269
- [Result] Koo BK, Um SH, Seo DS, Joo SK, Bae JM, Park JH, Chang MS, Kim JH, Lee J, Jeong WI, Kim W. Growth differentiation factor 15 predicts advanced fibrosis in biopsy-proven non-alcoholic fatty liver disease. Liver Int. 2018 Apr;38(4):695-705. doi: 10.1111/liv.13587. Epub 2017 Sep 30. PMID 28898507
- [Result] Joo SK, Kim W, Kim D, Kim JH, Oh S, Lee KL, Chang MS, Jung YJ, So YH, Lee MS, Bae JM, Kim BG. Steatosis severity affects the diagnostic performances of noninvasive fibrosis tests in nonalcoholic fatty liver disease. Liver Int. 2018 Feb;38(2):331-341. doi: 10.1111/liv.13549. Epub 2017 Sep 5. PMID 28796410
- [Result] Kim D, Kim W, Joo SK, Bae JM, Kim JH, Ahmed A. Subclinical Hypothyroidism and Low-Normal Thyroid Function Are Associated With Nonalcoholic Steatohepatitis and Fibrosis. Clin Gastroenterol Hepatol. 2018 Jan;16(1):123-131.e1. doi: 10.1016/j.cgh.2017.08.014. Epub 2017 Aug 18. PMID 28823829
- [Result] Kim JY, Park KJ, Hwang JY, Kim GH, Lee D, Lee YJ, Song EH, Yoo MG, Kim BJ, Suh YH, Roh GS, Gao B, Kim W, Kim WH. Activating transcription factor 3 is a target molecule linking hepatic steatosis to impaired glucose homeostasis. J Hepatol. 2017 Aug;67(2):349-359. doi: 10.1016/j.jhep.2017.03.023. Epub 2017 Mar 30. PMID 28365312
- [Result] Koo BK, Kim D, Joo SK, Kim JH, Chang MS, Kim BG, Lee KL, Kim W. Sarcopenia is an independent risk factor for non-alcoholic steatohepatitis and significant fibrosis. J Hepatol. 2017 Jan;66(1):123-131. doi: 10.1016/j.jhep.2016.08.019. Epub 2016 Sep 4. PMID 27599824
- [Result] Lee MS, Bae JM, Joo SK, Woo H, Lee DH, Jung YJ, Kim BG, Lee KL, Kim W. Prospective comparison among transient elastography, supersonic shear imaging, and ARFI imaging for predicting fibrosis in nonalcoholic fatty liver disease. PLoS One. 2017 Nov 27;12(11):e0188321. doi: 10.1371/journal.pone.0188321. eCollection 2017. PMID 29176844
- [Derived] Lee DH, Sung SU, Lee YK, Lim IH, Jang H, Joo SK, Park JH, Chang MS, So YH, Kim W; Innovative Target Exploration of NAFLD (ITEN) Consortium. A sequential approach using the age-adjusted fibrosis-4 index and vibration-controlled transient elastography to detect advanced fibrosis in Korean patients with non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2022 Apr;55(8):994-1007. doi: 10.1111/apt.16766. Epub 2022 Jan 9. PMID 35005800
- [Derived] Kim D, Kim W, Joo SK, Han J, Kim JH, Harrison SA, Younossi ZM, Ahmed A. Association between body size-metabolic phenotype and nonalcoholic steatohepatitis and significant fibrosis. J Gastroenterol. 2020 Mar;55(3):330-341. doi: 10.1007/s00535-019-01628-z. Epub 2019 Sep 18. PMID 31535207
- [Derived] Kim D, Kim W, Joo SK, Kim JH, Harrison SA, Younossi ZM, Ahmed A. Predictors of nonalcoholic steatohepatitis and significant fibrosis in non-obese nonalcoholic fatty liver disease. Liver Int. 2019 Feb;39(2):332-341. doi: 10.1111/liv.13983. Epub 2018 Oct 27. PMID 30298568